CLINICAL TRIAL: NCT03214146
Title: An Open-label, Phase 1 Trial for Safety and Efficacy Study of 2nd Cycle Treatment After 6 Months of 1st Cycle HLA-haplo Matched Allogenic Bone Marrow Derived Stem Cell("HYNR-CS-Allo Inj") Treatment in Amyotrophic Lateral Sclerosis(ALS)
Brief Title: Safety/Efficacy Study of 2nd Cycle Treatment After 6 Months of 1st Cycle HLA-haplo Matched Allogenic Bone Marrow Derived Stem Cell Treatment in ALS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hanyang University Seoul Hospital (Other)
Collaborators: Corestemchemon, Inc. (Industry)
Responsible Party: Principal Investigator, Seung Hyun Kim, Principal Investigator, Hanyang University Seoul Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYNR-CS-Allo-02
Record Dates: First submitted 2017-07-09; First posted 2017-07-11 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Motor Neuron Disease; Neuromuscular Disease; Neurodegenerative Disease; Central Nervous System Disease; HLA-haplo matched allogenic bone marrow derived stem cells
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Neuromuscular Diseases; Neurodegenerative Diseases; Central Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HYNRCS-Allo inj. (Experimental): 2 cycles of HYNRCS-Allo inj. with 6 months interval through intrathecal injection.
  *1 cycle of HYNRCS-Allo inj. is 2 times administration with 28 days interval by intrathecal.
  Interventions: Biological: HYNRCS-Allo inj

INTERVENTIONS:
Biological: HYNRCS-Allo inj — The patients enrolled in the trial will be successively allocated into single cohort for HYNRCS-Allo inj., 1.0 X 10^6 cells/kg according to the protocol design.
  Other Names: HLA-haplo Matched Allogenic Bone Marrow Derived Stem Cell

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of HLA-haplo matched Allogenic Bone Marrow Derived stem cells("HYNRCS-Allo-ALS-02 inj"), through intrathecal delivery for the repeated treatment after 6 months of first treatment in patients with amyotrophic lateral sclerosis(ALS).

This study is an open label, single-dose study to assess the safety and efficacy of HLA-haplo matched Allogenic Bone Marrow Derived stem cells("HYNRCS-Allo-ALS-02 inj")

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis is a progressive neurodegenerative disease characterized by motor neuron loss. Despite of many trials for disease-modifying, no treatment has so far changed natural course of disease.

The investigators had performed the pre-clinical and clinical studies using autologous bone marrow-derived stem cells in ALS. In the investigators' results of clinical trial, intrathecal injection of autologous bone marrow-derived stem cells is safe and could slow down disease progression and might be used as a disease modifying strategy in patients with ALS.

In the new field, like cell therapy, it is an important issue whether a bone marrow derived mesenchymal stem cells can be used as an allograft. Many investigators had showed that the immunoprivileged and immunosuppressive properties of mesenchymal stem cells result from the absence of major histocompatibility class II antigens and the secretion of T helper type 2 cytokines.

One potential advantage of allogenic bone marrow derived cells could be avoiding the need for procedural delay before treatment. And it is also hypothesized that the function of autologous bone marrow derived cells could be impaired in patients with co-morbidities or advanced age.

This study is to evaluate safety and efficacy of repeated treatment after 6 months of first HYNRCS-Allo-ALS-02 inj(HLA-haplo matched Allogenic bone marrow-derived stem cells) treatment in patients with ALS.

The patients enrolled in the trial will be successively allocated into single cohort for HYNRCS-Allo-ALS-02 inj., 1.0 X 10^6 cells/kg, according to the protocol design. Only a maximum of six patients will be given a particular dosage.

The scheduled assessments and visits will be carried out over three periods: run-in period, treatment period, and follow-up period.

The run-in period includes the screening visit where a written informed consent is obtained and the screening period where patients are assessed for eligibility. It will be completed within 56 days prior to enrollment. The patients meeting inclusion criteria will start the treatment period.

During the treatment period, subjects will be administered HYNRCS-Allo-ALS-02 inj. 2 times(first treatment) by intrathecal administration with 28 days interval and there will be repeated treatment after 6 months of the first treatment.

The Follow-up period starts once subjects complete the treatment period and will continue until the final follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 25 and 80 years old
* Patients diagnosed as 'Possible with lab-supported' or 'Possible' or 'Probable' or 'Definite' ALS according to the World Federation of Neurology El Escorial criteria
* Patients whose duration of disease is within 5 years from the first diagnosis
* Patients with ALSFRS-R score within 21 to 46 at screening
* Patients who can visit to a hospital by walk personally or by protector's help
* Patients who provide the written consent by oneself or his/her legal representative
* Patients who has HLA-haplo matched Bone marrow donor

Exclusion Criteria:

* Patients who doesn't appropriate to the diagnostic criteria of ALS
* Patients who doesn't have HLA-haplo-matched bone marrow donor
* Patients suspected of adverse effect after stem cell injection(patients suspected of malignant tumor, risk group of psychogenic shock, patients with serious hypertension)
* Patients with ALSFRS-R score below 21 at screening
* Patients performed Tracheostomy at screening
* Patients with suspected 20% or less of Forced vital capacity(FVC) at screening
* Patients who doesn't agree with written consent form by oneself of his/her legal representative
* Patients who have taken any other drug for clinical trial within the past 3 months at screening entry
* Patients with epilepsy
* Patients with severe medical disease
* Pregnant woman, lactating woman, female patients who has a pregnancy planning or who doesn't agree with adoption of contraception methods proper medically, male patients who doesn't agree with adoption of contraception methods proper to his partner during participating this study
* Patients with hemorrhagic tendency at screening
* Patients with a known history of hypersensitivity/allergy to penicillin and streptomycin
* Patients with severe psychotic diseases (such as alzheimer, schizophrenia excepts slight cognitive dysfunction and secondary emotional disorder)

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
The Incidence of any treatment related serious adverse events(SAE) | 12 months

SECONDARY OUTCOMES:
ALS-Functional rating scales(ALS-FRS) | 12 months
Incidence & Degree of Adverse Events(AE) | 12 months
PRA test to identify generation status of HLA antibody | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Seung Hyun Kim, M.D.,Ph.D., Principal Investigator — Hanyang University
Locations (1):
- Hanyang University Seoul Hospital, Cell Therapy Center for Neurologic Disorders, Seoul, Haengdang-dong, Seongdong-gu, South Korea

IPD SHARING:
Plan to Share IPD: No